CLINICAL TRIAL: NCT03858400
Title: Electrophysiological Responses to External Stimuli of Patients Evaluated as Unconscious Patient in Critical Care Units: Preliminary Results of 10 Patients
Brief Title: Electrophysiological Tests on Unconscious Patient
Status: Completed | Type: Observational
Sponsor: Nevsehir Public Hospital (Other Government)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/407
Record Dates: First submitted 2019-02-27; First posted 2019-02-28 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Conditions of Brain
Keywords: Unconscious patient; critical care unit; electrophysiological test
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most patients with minimal consciousness status in Critical Care Units (CCU) are considered as an 'unconscious patient' with a neurological examination. Evaluating these patients as unconscious patients may lead to neglect of psychosocial needs in patient-care, a continuation of unchanged treatment protocols for a long time and desperate evaluation of prognosis. In this study, the investigators aimed to evaluate the emotional responses of patients who were considered by the healthcare providers and relatives of patients as an 'unconscious patient' by using electrophysiological tests.

DETAILED DESCRIPTION:
Most patients with minimal consciousness status in Critical Care Units (CCU) are considered as an 'unconscious patient' with a neurological examination. A study showed that only 5% of intensive care nurses communicate with the unconscious patients and the content of the communication with them is to explain only the procedures to apply. Lack of communication with these patients can be transformed into the sense of 'non-responsive patient' among healthcare providers. Evaluating these patients as unconscious patients may lead to neglect of psychosocial needs in patient-care, a continuation of unchanged treatment protocols for a long time and desperate evaluation of prognosis. Moreover, it may lead to burnout syndrome over time for physicians and nurses in the CCU. In particular, the futile care perception of caregiving about unconscious patient prolongs the recovery process and length of stay in CCU. On the other hand, it may lead to the occupation of beds and increases the costs. Coma and sedation scoring systems such as Glasgow Coma Scale (GCS), Ramsey Sedation Scale (RSS) and Full Outline of Unresponsiveness (FOUR) have traditionally been used to assess the consciousness in CCU. These scoring systems may be insufficient to assess the psychophysiological status of the patients. Some researches on the unconscious patients have shown that these patients are aware of their surroundings. However, the data for these studies were obtained from interviews with patients who were previously experiencing unconsciousness, or with caregivers in CCU. The balance between sympathetic and parasympathetic systems is controlled by the autonomic nervous system. The response of the sympathetic system to external stimuli is different in many organs of the body. For example, a painful stimulus causes myosis in the eyes, hypertension, and tachycardia. Emotional stimuli also activate the sympathetic system. Fear and excitement lead to mydriasis, elevation of blood pressure and tachycardia, and activation of eccrine gland increase to release of sweating. Electrophysiological tests are objective methods in which the physiological signals and psychological states of emotion are acquired by noninvasively connected superficial electrodes. Through this method, the R-R interval (velocity analysis) can be evaluated by the Poincare Plot analysis in the electrocardiogram (ECG) to measure the electrical activity of the heart. Electrooculography (EOG) is a test that evaluates the eyes movements. In EOG, the source of the signals is the stationary electrical potential between the cornea and the retina. The EOG is composed of the changes of the electricity based on the movements of the eyeball around the eye center. Galvanic skin response (GSR) is a test used to measure skin conductivity and reflects electrodermal activity. In addition, blood pressure and pulse rate (PR) measurements provide information about the psychophysiological status of patients as a result of a sympathetic activity. In this study, the investigators aimed to evaluate the emotional responses of patients who were considered by the healthcare providers and relatives of patients as an 'unconscious patient' by using electrophysiological tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GCS score of 3,
* GCS score of 4 or 5 only when their motor response is 2 or 3,
* ≥18 years of age

Exclusion Criteria:

* Patients with GCS score ≥6,
* taking medication for sedation,
* motor neuron diseases such as ALS,
* suspected or actual brain death
* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who be considered to be unconscious in our CCU's
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Electrophysiological evaluating | 40 minutes
  To detect electrophysiologically that patients who were thought to be unconscious were responsive to the external stimuli of health providers and relatives.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akif Yazar, MD, Study Director — Nevsehir Public Hospital
Locations (1):
- Mehmet Akif YAZAR, Nevşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wieser M, Buetler L, Koenig A, Riener R. Quantitative description of the state of awareness of patients in vegetative and minimally conscious state. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:5533-6. doi: 10.1109/IEMBS.2010.5626763. PMID 21096471
- [Result] Schnakers C, Vanhaudenhuyse A, Giacino J, Ventura M, Boly M, Majerus S, Moonen G, Laureys S. Diagnostic accuracy of the vegetative and minimally conscious state: clinical consensus versus standardized neurobehavioral assessment. BMC Neurol. 2009 Jul 21;9:35. doi: 10.1186/1471-2377-9-35. PMID 19622138